CLINICAL TRIAL: NCT07316803
Title: Study on the Effectiveness of a Group Intervention on Romantic Relationships in Young Adults With Severe Mental Illness
Brief Title: Group Intervention for Romantic Relationships in Young Adults With Severe Mental Illness
Acronym: A2C'estMieuxVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de Ville-Evrard, France (Other)
Responsible Party: Principal Investigator, Raluca ROSETTI, Principal Investigator, Centre hospitalier de Ville-Evrard, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLER 02 - 001_A2 C'estMieux VE
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Severe Mental Illness; Schizophrenia; Bipolar Disorder; Major Depressive Disorder
Keywords: severe mental illness; omantic relationships; intimate relationships; social functioning; loneliness; self-esteem; self-stigma; recovery; group intervention; psychosocial intervention; social skills training; relationship skills; mental health rehabilitation; adults with mental illness
MeSH Terms: conditions — Mental Disorders; Schizophrenia; Bipolar Disorder; Depressive Disorder, Major; Social Adjustment

STUDY DESIGN:
Intervention Model Description: This study uses a repeated single-case experimental design in which all participants receive the same group-based intervention. Participants serve as their own control, with outcomes measured before the intervention, immediately after completion of the 12-session program, and at a three-month follow-up.
Masking Description: This is an open-label study. Participants and study staff are aware of the intervention being delivered. Masking is not feasible due to the behavioral and group-based nature of the intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- À deux, c'est mieux Group Intervention (Experimental): Participants receive the "À deux, c'est mieux" group-based psychosocial intervention, a structured program designed to improve romantic and social relationship functioning in adults living with a severe mental illness. The intervention is delivered in small groups over 12 weekly sessions led by trained mental health professionals.
  Interventions: Behavioral: À deux, c'est mieux (Better Together) Group Intervention

INTERVENTIONS:
Behavioral: À deux, c'est mieux (Better Together) Group Intervention — The "À deux, c'est mieux" intervention is a manualized, group-based psychosocial program consisting of 12 weekly sessions. The program targets the development of romantic relationship skills, including communication, emotional regulation, social cognition, and intimacy-related behaviors. Sessions follow a progressive structure, beginning with relationship initiation and communication skills and gradually addressing more sensitive topics such as emotional intimacy, attachment-related anxiety, and sexuality. The intervention is inclusive of sexual and gender diversity and is delivered by trained mental health professionals in groups of 4 to 6 participants.
  Other Names: Better Together

SUMMARY:
This study evaluates a group-based intervention designed to improve romantic and social relationship skills in adults living with a severe mental illness (SMI), such as schizophrenia, bipolar disorder, or major depressive disorder.

Many adults with SMI experience loneliness, social isolation, and difficulties forming romantic relationships, even though most express a strong desire for intimacy. These challenges may be related to social skill difficulties, stigma, low self-esteem, and limited opportunities to develop healthy relationships.

The "À deux, c'est mieux" (Better Together) program is a structured 12-session group intervention focused on developing communication skills, emotional regulation, social understanding, and healthy romantic relationship behaviors. Sessions are led by trained mental health professionals and take place in small groups.

Participants will complete assessments before starting the program, at the end of the 12 sessions, and three months later. The study will examine changes in romantic relationship skills, quality of life, loneliness, self-esteem, self-stigma, and recovery.

The purpose of this study is to determine whether this intervention improves romantic and social functioning and overall well-being, and whether it is acceptable and relevant for adults living with severe mental illness.

DETAILED DESCRIPTION:
This multicenter, prospective study examines the effects of the "À deux, c'est mieux" group intervention on romantic and social functioning in adults living with a severe mental illness (SMI).

Romantic relationships are an important component of emotional well-being and social integration. However, adults with SMI often face significant barriers to forming and maintaining intimate relationships, including social skill challenges, limited social networks, stigma, low self-esteem, and fear of rejection. Although most express a desire for romantic relationships, many feel unprepared to develop or sustain healthy partnerships.

The "À deux, c'est mieux" program is a manualized group intervention consisting of 12 weekly sessions. The program follows a progressive structure, beginning with topics such as attraction, communication, and relationship initiation, and gradually addressing more sensitive themes including emotional intimacy, attachment-related anxiety, and sexuality. The intervention uses group discussions, experiential exercises, and practical strategies to promote healthy romantic relationship skills, emotional awareness, and social cognition. The program is inclusive of sexual and gender diversity.

The intervention will be delivered in small groups of 4 to 6 participants by trained mental health professionals. Outcomes will be assessed at three time points: before the intervention (baseline), immediately after completion of the 12 sessions, and at a three-month follow-up. The study uses a repeated single-case experimental design in which each participant serves as their own control, allowing for comparison of outcomes over time without the use of an inactive control group.

The primary outcome is improvement in romantic relationship functioning. Secondary outcomes include quality of life, perceived loneliness, self-esteem, internalized stigma, and recovery. Data will be analyzed using repeated-measures statistical methods to evaluate changes across assessment time points.

This study addresses an important gap in mental health care by focusing on romantic relationships and intimacy, areas that are often overlooked but central to recovery and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older
* Diagnosis of a severe mental illness (e.g., schizophrenia, bipolar disorder, or major depressive disorder)
* Currently single
* Motivated to improve romantic and social relationships and to pursue a romantic relationship
* Received mental health care within the past two years
* Able and willing to provide informed consent

Exclusion Criteria:

* Inability to speak or read French
* Currently receiving acute or crisis-level psychiatric care
* Unable to comply with study procedures or group rules (e.g., maintaining sobriety during sessions)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-11-03 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in Romantic Relationship Functioning | Baseline (pre-intervention), end of the 12-session intervention, and 3-month follow-up
  Romantic relationship functioning will be assessed using the Romantic Relationships Functioning Scale, a self-report questionnaire measuring skills related to initiating, maintaining, and experiencing healthy romantic relationships. Higher scores indicate better romantic relationship functioning.

SECONDARY OUTCOMES:
Change in Quality of Life | Baseline, end of the 12-session intervention, and 3-month follow-up
  Quality of life will be measured using the Schizophrenia Quality of Life Questionnaire (SQOL-18), a self-report scale assessing psychological well-being, self-esteem, family relationships, and social functioning. Higher scores indicate better quality of life.
Change in Perceived Loneliness | Baseline, end of the 12-session intervention, and 3-month follow-up
  Perceived loneliness will be assessed using the UCLA Loneliness Scale (ULS-8), a self-report measure evaluating subjective feelings of loneliness and social isolation. Higher scores indicate greater loneliness.
Change in Self-Esteem | Baseline, end of the 12-session intervention, and 3-month follow-up
  Self-esteem will be assessed using the Self-Esteem Rating Scale (SERS), a self-report questionnaire measuring positive and negative self-evaluations. Higher scores indicate higher self-esteem.
Change in Internalized Stigma | Baseline, end of the 12-session intervention, and 3-month follow-up
  Internalized stigma will be measured using the Internalized Stigma of Mental Illness Scale (ISMI), a self-report questionnaire assessing self-stigma related to mental illness. Higher scores indicate greater internalized stigma.
Change in Recovery | Baseline, end of the 12-session intervention, and 3-month follow-up
  Recovery will be assessed using the Stages of Recovery Instrument (STORI), a self-report measure evaluating subjective recovery processes in individuals with mental illness.

CONTACTS AND LOCATIONS:
Overall Officials: Raluca ROSETTI, Principal Investigator, Principal Investigator — Psychiatrist, EPS Ville-Evrard
Locations (2):
- France (2):
  - HDJ (Hôpital de Jour), Épinay-sur-Seine, Île-de-France Region
  - L'UNIRRE (Unité Référente de Réhabilitation), Neuilly-sur-Marne, Île-de-France Region

REFERENCES:
- [Background] White R, Haddock G, Campodonico C, Haarmans M, Varese F. The influence of romantic relationships on mental wellbeing for people who experience psychosis: A systematic review. Clin Psychol Rev. 2021 Jun;86:102022. doi: 10.1016/j.cpr.2021.102022. Epub 2021 Mar 20. PMID 33819779
- [Background] Weissbourd et al. The Talk: How Adults Can Promote Young People's Healthy Relationships and Prevent Misogyny and Sexual Harassment. (Harvard School of Education, 2017)
- [Background] Pillay R, Lecomte T, Abdel-Baki A. Factors limiting romantic relationship formation for individuals with early psychosis. Early Interv Psychiatry. 2018 Aug;12(4):645-651. doi: 10.1111/eip.12353. Epub 2016 May 17. PMID 27186857
- [Background] Macdonald EM, Hayes RL, Baglioni AJ Jr. The quantity and quality of the social networks of young people with early psychosis compared with closely matched controls. Schizophr Res. 2000 Nov 30;46(1):25-30. doi: 10.1016/s0920-9964(00)00024-4. PMID 11099882
- [Background] Hache-Labelle C, Abdel-Baki A, Lepage M, Laurin AS, Guillou A, Francoeur A, Bergeron S, Lecomte T. Romantic relationship group intervention for men with early psychosis: A feasibility, acceptability and potential impact pilot study. Early Interv Psychiatry. 2021 Aug;15(4):753-761. doi: 10.1111/eip.13012. Epub 2020 Jun 23. PMID 32578401
- [Background] Bonfils KA, Firmin RL, Salyers MP, Wright ER. Sexuality and intimacy among people living with serious mental illnesses: Factors contributing to sexual activity. Psychiatr Rehabil J. 2015 Sep;38(3):249-55. doi: 10.1037/prj0000117. Epub 2015 Feb 9. PMID 25664756
- [Background] Cloutier B, Lecomte T, Diotte F, Lamontagne J, Abdel-Baki A, Daneault JG, Gelineau Rabbath ME, de Connor A, Perrine C. Improving Romantic Relationship Functioning Among Young Men With First-Episode Psychosis: Impact of a Novel Group Intervention. Behav Modif. 2023 Sep;47(5):1170-1192. doi: 10.1177/01454455231186586. Epub 2023 Jul 26. PMID 37496322
- [Background] Borge L, Martinsen EW, Ruud T, Watne O, Friis S. Quality of life, loneliness, and social contact among long-term psychiatric patients. Psychiatr Serv. 1999 Jan;50(1):81-4. doi: 10.1176/ps.50.1.81. PMID 9890584
- [Background] Beyers W, Seiffge-Krenke I. Does Identity Precede Intimacy? Testing Erikson's Theory on Romantic Development in Emerging Adults of the 21st Century. Journal of Adolescent Research. 2010;25(3):387-415.